CLINICAL TRIAL: NCT05425459
Title: Re-Evaluation of the Corvia Atrial Shunt Device in a Precision Medicine Trial to Determine Efficacy in Mildly Reduced or Preserved Ejection Fraction (EF) Heart Failure (Protocol #2201)
Brief Title: RESPONDER-HF Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2201
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Heart Failure, Diastolic
Keywords: Heart failure with preserved ejection fraction (HFpEF); Heart failure with midrange ejection fraction (HFmrEF); Interatrial Shunt
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — Ice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Participants randomized to the treatment arm will undergo a fluoroscopic and intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) guided trans-septal puncture and InterAtrial Shunt Device (IASD) System II implant procedure.
  Interventions: Device: Corvia Atrial Shunt System / IASD System II
- Control (Sham Comparator): Participants randomized to the control arm will undergo fluoroscopy and intracardiac echocardiography from the femoral vein or transesophageal echocardiography, for examination of the atrial septum and left atrial appendage.
  Interventions: Other: Intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE)

INTERVENTIONS:
Device: Corvia Atrial Shunt System / IASD System II — The primary component of the system is an implant placed in the atrial septum designed to allow left to right flow between the left atrium and right atrium to reduce the elevated left atrial pressure.
  Arms: Treatment
Other: Intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) — Intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) for examination of the atrial septum and left atrium.
  Arms: Control

SUMMARY:
Multicenter, Prospective, Randomized, Sham Controlled, Double Blinded Clinical Trial, with; 1:1 randomization

DETAILED DESCRIPTION:
Following supine bicycle exercise hemodynamic assessment to verify eligibility, patients are sedated then randomized to the treatment or control group. Patients in both arms will undergo placement of femoral venous access sheath.

Patients randomized to the treatment arm will undergo a fluoroscopically and intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) guided trans-septal puncture and Corvia Atrial Shunt implant procedure. Patients randomized to the control arm will undergo ICE from the femoral vein or TEE for examination of the atrial septum and left atrium.

Patients will be evaluated at pre-specified time intervals and followed for 5 years.

All patients will be unblinded after the 24 month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic symptomatic heart failure (HF) documented by the following:

   1. Symptoms of HF requiring current treatment with diuretics if tolerated for ≥ 30 days AND
   2. New York Heart Association (NYHA) class II; OR NYHA class III, or ambulatory NYHA class IV symptoms; AND
   3. ≥ 1 HF hospital admission (with HF as the primary, or secondary diagnosis); or treatment with intravenous (IV) diuretics; or intensification of oral diuresis within the 12 months prior to study entry; OR an NT-proB-type Natriuretic Peptide (NT-pro BNP) value > 150 pg/ml in normal sinus rhythm, > 450 pg/ml in atrial fibrillation, or a brain natriuretic peptide (BNP) value > 50 pg/ml in normal sinus rhythm, > 150 pg/ml in atrial fibrillation within the past 6 months
2. Ongoing stable guideline-directed medical therapy (GDMT) HF management and management of comorbidities according to the 2022 American College of Cardiology (ACC)/American Heart Association (AHA) Guidelines for the Management of Heart Failure. Stable management includes a minimum period of 4 weeks post-hospitalization for any cause, including treatment with IV diuretics
3. Site determined echocardiographic LV ejection fraction ≥ 40% within the past 6 months, without documented ejection fraction < 30% in the 5 years prior.
4. Site determined echocardiographic evidence of diastolic dysfunction documented by one or more of the following:

   1. Left Atrial (LA) diameter > 4 cm; or
   2. Diastolic LA volume > 50 or LA volume index > 28 ml/m2 or
   3. Lateral e' < 10 cm/s; or
   4. e' < 8 cm/s; or
5. Site determined elevated pulmonary capillary wedge pressure (PCWP) with a gradient compared to right atrial pressure (RAP) documented by end-expiratory PCWP during supine ergometer exercise ≥ 25 millimeters of mercury (mm Hg), and greater than RAP by ≥ 5 mm Hg.
6. Resting RAP ≤ 14 mmHg
7. Site determined hemodynamic evidence of peak exercise pulmonary vascular resistance (PVR) < 1.75 Wood units
8. Age ≥ 40 years old
9. Participant has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the Institutional Review Board (IRB) or Ethics Committee (EC)
10. Participant is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams
11. Transseptal catheterization and femoral vein access to the right atrium is determined to be feasible by site interventional cardiology investigator.

Exclusion Criteria:

1. Advanced heart failure defined as one or more of the below:

   1. ACC/AHA/European Society of Cardiology (ESC) Stage D heart failure, non-ambulatory NYHA Class IV HF
   2. Cardiac index < 2.0 L/min/m2
   3. Inotropic infusion (continuous or intermittent) for EF < 40% within the past 6 months
   4. Patient is on the cardiac transplant waiting list.
2. Inability to perform 6-minute walk test (distance < 50 meters), OR 6-minute walk test > 600m
3. The patient has verified that the ability to walk 6 minutes is limited primarily by joint, foot, leg, hip or back pain; unsteadiness or dizziness or lifestyle (and not by shortness of breath and/or fatigue and/or chest pain)
4. Right ventricular dysfunction, assessed by the site cardiologist and defined as one or more of the following:

   1. More than mild right ventricular (RV) dysfunction as estimated by transthoracic echocardiogram (TTE); OR
   2. TAPSE < 1.4 cm; OR
   3. Right ventricular (RV) size ≥ left ventricular (LV) size as estimated by TTE; OR
   4. Ultrasound or clinical evidence of congestive hepatopathy; OR
   5. Evidence of RV dysfunction defined by TTE as an RV fractional area change < 35%.
5. Any implanted cardiac rhythm device
6. Structural heart repair aortic valve replacement (AVR) or mitral valve replacement (MVR) (surgical or percutaneous) within the past 12 months; planned valve intervention in the next 3 months, or presence of hemodynamically significant valve disease as assessed by the site cardiologist and defined as:

   1. Mitral valve disease grade ≥ 3+ mitral regurgitation (MR) or > mild Mitral Stenosis (MS); OR
   2. Tricuspid valve (TR) regurgitation grade ≥ 2+ TR; OR
   3. Aortic valve disease ≥ 2+ aortic regurgitation (AR) or > moderate aortic stenosis (AS)
7. Echocardiographic evidence of intra-cardiac mass, thrombus or vegetation
8. Participants with existing or surgically closed (with a patch) atrial septal defects. Participants with a patent foramen ovale (PFO), who meet PCWP criteria despite the PFO, are not excluded
9. Myocardial Infarction (MI) and/or percutaneous cardiac intervention within past 3 months; Coronary Artery Bypass Graft (CABG) surgery in past 3 months or any planned cardiac interventions in the 3 months following enrollment.
10. Known clinically significant un-revascularized coronary artery disease, defined as: coronary artery stenosis with angina or other evidence of ongoing active coronary ischemia
11. Known clinically significant untreated carotid artery stenosis likely to require intervention
12. Atrial fibrillation with resting heart rate (HR) > 100 beats-per-minute (BPM)
13. Hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, cardiac amyloidosis or infiltrative cardiomyopathy (e.g. hemochromatosis, sarcoidosis)
14. History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 6 months
15. Participant is contraindicated to receive either dual antiplatelet therapy, or an oral anticoagulant; or has a documented coagulopathy
16. Anemia with Hemoglobin < 10 g/dl
17. Chronic pulmonary disease requiring continuous home oxygen, OR significant chronic pulmonary disease defined as forced expiratory volume (FEV)1 <1Liter
18. Resting arterial oxygen saturation < 95% on room air, <93% when residing at high altitude
19. Currently requiring dialysis; or estimated glomerular filtration rate eGFR < 25ml/min/1.73 m2 by chronic kidney disease (CKD) CKD-Epi equation
20. Systolic blood pressure > 170 mm Hg at screening
21. Significant hepatic impairment defined as 3 times upper limit of normal of transaminases, total bilirubin, or alkaline phosphatase
22. Participants on significant immunosuppressive treatment or on systemic steroid treatment
23. Life expectancy less than 12 months for known non-cardiovascular reasons
24. Known hypersensitivity to nickel or titanium
25. Women of childbearing potential
26. Severe obstructive sleep apnea not treated with continuous positive airway pressure (CPAP) or other measures
27. Body Mass Index (BMI) > 45; BMI 40 - 45 is also excluded unless in the opinion of the investigator, vascular access can be obtained safely
28. Severe depression and/or anxiety
29. Currently participating in an investigational drug or device study that would interfere with the conduct or results of this study. Note: trials requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational
30. In the opinion of the investigator, the Participant is not an appropriate candidate for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Endpoint | Up to 12 months
  The primary endpoint is a composite of heart failure event rates and Kansas City Cardiomyopathy Questionnaire (KCCQ) at 12 months.
  Responses are given on a Likert scale that for each individual item is scored on a scale of 0-100 with higher scores indicating better health.

SECONDARY OUTCOMES:
The incidence of cardiovascular mortality | Up to 12 months
  The incidence of cardiovascular mortality through 12 months.
The rate of time-to-cardiovascular mortality | Up to 12 months
  Time-to-cardiovascular mortality through 12 months.
The rate of major adverse cardiac periprocedural events | Through 30 days
  Major adverse cardiac periprocedural events through 30 days defined as:
  1. Cardiac death
  2. Myocardial infarction
  3. Cardiac tamponade
  4. Emergency cardiac surgery.
The incidence of non-fatal, ischemic stroke | Through 12 months
  Incidence of non-fatal, ischemic stroke
The rate of new onset or worsening of kidney dysfunction | Through 12 months
  New onset or worsening of kidney dysfunction (defined as estimated glomerular filtration rate (eGFR) decrease of > 20 ml/min/1.73 m2) through 12 months
The incidence of thrombo-embolic complications including transient ischaemic attack (TIA) and systemic embolization) | Through 12 months
  The incidence of thrombo-embolic complications (TIA and systemic embolization) through 12 months
The incidence of newly acquired persistent or permanent atrial fibrillation (AF) or atrial flutter | Through 12 months
  The incidence of newly acquired persistent or permanent AF or atrial flutter
The incidence of participants with a ≥30% decrease in Tricuspid Annular Plane Systolic Excursion (TAPSE) | Through 12 months
  The incidence of participants with a ≥30% decrease Tricuspid Annular Plane Systolic Excursion (TAPSE)
The rate of heart failure (HF) admissions | Through 24 months
  Total rate (first plus recurrent) per patient year of heart failure (HF) admissions or healthcare facility visits for intravenous diuresis or urgent visits with intensification of oral diuresis for HF through 24 months, analyzed when the last randomized participant completes 12 months follow-up.
The change in New York Heart Association (NYHA) Class | 12 months
  Change in NYHA functional Class between baseline and 12 months
The change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Score | 12 months
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Score between baseline and 12 months, categorized as proportion of patients with changes of ≤0, >0 - 5, >5 - 10, >10 - 15, >15 - 20, >20 - 25, >25 points. Responses are given on a Likert scale that for each individual item is scored on a scale of 0-100 with higher scores indicating better health

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern Memorial Hospital; Martin Leon, MD, Principal Investigator — Columbia University
Locations (61):
- United States (33):
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - Christiana Care Health Services, Newark, Delaware
  - Memorial Regional Hospital, Hollywood, Florida
  - NCH Naples, Naples, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Northside Hospital Gwinnett Campus, Lawrenceville, Georgia
  - Wellstar Kennestone, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Endeavor Health-Northshore, Glenview, Illinois
  - LSU Health Shreveport, Shreveport, Louisiana
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - UMass Memorial Hospital University Campus, Worcester, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell, New York, New York
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinatti Medical Center, Cincinnati, Ohio
  - Cleveland Clinic OH, Cleveland, Ohio
  - Ohio State University Wexner medical Center, Columbus, Ohio
  - St. Francis Hospital (Heart Hospital), Tulsa, Oklahoma
  - OHSU Hospital, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Cardiovascular Institute (CVI) Research, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - North Central Heart-Avera, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee
  - Baylor St. Luke's Medical Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - West Virginia Heart and Vascular, Morgantown, West Virginia
- Australia (4):
  - St. Vincents Hospital, Darlinghurst, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- LKH University Clinic, Graz, Austria
- Onze-Lieve-Vrouwziekenhuis Aalst (OLV), Aalst, Belgium
- Canada (2):
  - St. Paul's Hospital Providence Health Care, Vancouver, British Columbia
  - Unity Health Toronto St. Michael's Hospital, Toronto, Ontario
- Germany (19):
  - University Heart Center Bad Krozingen, Bad Krozingen
  - Kerckhoff Klinik, Bad Nauheim
  - Hospital Charité - University Medicine Berlin, Berlin
  - Vivantes Clinic Friedrichshain Berlin, Berlin
  - DRK Clinics Berlin Koepenick, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - University Hospital Cologne, Cologne
  - Heart Center of Dresden, Dresden
  - UK Duesseldorf, Düsseldorf
  - University Heart Center Freiburg, Freiburg im Breisgau
  - Georg-August Universität Gottingen Universitätsklinikum Göttingen Klinik für Kardiologie und Pneumologie, Göttingen
  - Marienkrankenhaus Hospital Hamburg, Hamburg
  - Asklepios Clinic Altona Hamburg, Hamburg
  - Herzzentrum Leipzig - Universitätsklinik, Leipzig
  - University Hospital Schleswig-Holstein (UKSH) Luebeck, Lübeck
  - University Hospital Münster, Münster
  - Helios Kliniken Schwerin, Schwerin
  - Ulm University Hospital, Ulm
  - University Hospital Wurzburg, Würzburg
- UMCG - Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borlaug BA, Blair J, Bergmann MW, Bugger H, Burkhoff D, Bruch L, Celermajer DS, Claggett B, Cleland JGF, Cutlip DE, Dauber I, Eicher JC, Gao Q, Gorter TM, Gustafsson F, Hayward C, van der Heyden J, Hasenfuss G, Hummel SL, Kaye DM, Komtebedde J, Massaro JM, Mazurek JA, McKenzie S, Mehta SR, Petrie MC, Post MC, Nair A, Rieth A, Silvestry FE, Solomon SD, Trochu JN, Van Veldhuisen DJ, Westenfeld R, Leon MB, Shah SJ; REDUCE LAP-HF-II Investigators. Latent Pulmonary Vascular Disease May Alter the Response to Therapeutic Atrial Shunt Device in Heart Failure. Circulation. 2022 May 24;145(21):1592-1604. doi: 10.1161/CIRCULATIONAHA.122.059486. Epub 2022 Mar 31. PMID 35354306
- [Background] Shah SJ, Borlaug BA, Chung ES, Cutlip DE, Debonnaire P, Fail PS, Gao Q, Hasenfuss G, Kahwash R, Kaye DM, Litwin SE, Lurz P, Massaro JM, Mohan RC, Ricciardi MJ, Solomon SD, Sverdlov AL, Swarup V, van Veldhuisen DJ, Winkler S, Leon MB; REDUCE LAP-HF II investigators. Atrial shunt device for heart failure with preserved and mildly reduced ejection fraction (REDUCE LAP-HF II): a randomised, multicentre, blinded, sham-controlled trial. Lancet. 2022 Mar 19;399(10330):1130-1140. doi: 10.1016/S0140-6736(22)00016-2. Epub 2022 Feb 1. PMID 35120593